CLINICAL TRIAL: NCT01037504
Title: Phase I, Single Centre, Double-blind, Randomised, Placebo-controlled, Parallel-group Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Inhaled AZD5423 After Administration of Multiple Ascending Doses for 14 Days in Healthy Male and Female Subjects
Brief Title: AZD5423 Multiple Ascending Dose Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: D2340C00002; EudraCT No: 2009-016611-38
Record Dates: First submitted 2009-12-20; First posted 2009-12-23 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Healthy
Keywords: safety; tolerability; healthy; inhalation; Healthy volunteers
MeSH Terms: conditions — Respiratory Aspiration | interventions — 2,2,2-trifluoro-N-(1-((1-(4-fluorophenyl)-1H-indazol-5-yl)oxy)-1-(3-methoxyphenyl)-2-propanyl)acetamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Drug: AZD5423
  Interventions: Drug: AZD5423
- B (Placebo Comparator): Drug: Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD5423 — Suspension for nebulisation, inhaled. Each subject will receive an inhaled dose of AZD5423 or placebo once daily for 14 days. Starting dose as determined from SAD study and with up to 4 dose escalations not exceeding AstraZeneca pre-defined exposure limits.
  Arms: A
Drug: Placebo — Solution for nebulisation, inhaled. Each subject will receive an inhaled dose of AZD5423 or placebo once daily for 14 days.
  Arms: B

SUMMARY:
The aim of the study is to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of AZD5423 following multiple ascending dose administrations in healthy male and female subjects

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures
* Have a body mass index (BMI) between 18 and 30 kg/m2 and weigh at least 50 kg and no more than 100 kg

Exclusion Criteria:

* Any clinically significant disease or disorder
* Any clinically significant abnormalities at screening examination
* Use of any prescribed or non-prescribed medication

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Safety variables: adverse events | Assessment taken at screening visit, defined timepoints pre-dose and post-dose during treatment periods and follow-up visit. Volunteers will be monitored throughout the study for adverse events.

SECONDARY OUTCOMES:
Pharmacokinetics profile: concentration of AZD5423 in plasma | Samples taken at defined timepoints pre-dose and post-dose during treatment periods. Samples taken at approx. 39 timepoints.
Investigation of PD effects | Samples taken at screening visit, defined timepoints pre-dose and post-dose during treatment periods and follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Darren Wilbraham, Principal Investigator — Quintiles Drug Research Unit at Guy's Hospital, London, UK; Jorup Carin, Study Director — AstraZeneca R&D, Lund, Sweden
Locations (1):
- Research Site, London Bridge, Greater London, United Kingdom

REFERENCES:
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1255&filename=D2340C00002.pdf